CLINICAL TRIAL: NCT07293676
Title: The Effects of Instrument-Assisted Soft Tissue Mobilization and Vibration Therapy on Pain, Functionality, and Kinesiophobia in Individuals With Lumbar Disc Herniation
Brief Title: IASTM and Vibration Effects on Pain, Functionality, and Kinesiophobia in Lumbar Disc Herniation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-1887
Record Dates: First submitted 2025-12-02; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Vibration; Lumbar Disc Herniation; Soft Tissue Mobilization
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional exercise group (Active Comparator): The exercise program will be performed at home for four weeks, twice daily. Exercise progression will begin with 10 repetitions and will be individualized according to each participant's condition. Exercises that provoke pain will be discontinued as advised. Participants will be provided with an illustrated exercise brochure, and follow-up will be conducted once a week through phone calls.
  First, participants will be instructed to lie on their backs on a flat surface with their knees bent, placing approximately a 30 cm elevation (such as two pillows) under the calves to assume a relaxation position and maintain it for 30 seconds. The exercise program will include hip flexor and lumbar extensor stretching, hamstring stretching, bridge exercises, erector spinae strengthening (prone superman), quadruped alternating arm-leg raises, and cat-camel exercises.
  Interventions: Other: Exercise
- IASTM Group (Experimental): Instrument-assisted soft tissue mobilization treatment will be applied twice per week for a total of eight sessions. The intervention will be performed using stainless-steel tools of various sizes specifically designed for different anatomical regions (Figure 2). Instrument-assisted soft tissue mobilization will be administered to the iliocostalis lumborum, erector spinae, and quadratus lumborum muscles, as well as to the superficial and deep fascia. Before the application, a thin layer of petroleum jelly will be applied to the area to facilitate smooth gliding of the instrument.
  The IASTM treatment will be delivered for a total of six minutes, with each technique (sweep, fan, brush, and sweep) being performed for 8-10 repetitions along the affected muscle fibers.
  Interventions: Other: Exercise; Other: IASTM
- Percussion Massage Therapy Group (Experimental): Vibration massage therapy will be applied twice per week for a total of eight sessions. After positioning the participant in the prone position, the session will begin. For vibration massage, the No. 2 standard ball attachment of the Theragun™ and the Theragun Pro device, which provides 1750 percussions per minute, will be used. The Theragun will be held perpendicular to the muscle at all times, and no additional pressure other than the weight of the device itself will be applied. Throughout the procedure, the massage gun will be kept in continuous contact with the skin, maintaining consistent pressure.
  The vibration massage will be administered to the erector spinae and lumbar paravertebral muscle groups. A total of 10 minutes of percussion massage will be applied to the lateral portions of the lower back erector spinae muscles (5 minutes on each side), and the massage gun will be moved in a straight line from the distal to the proximal direction within approximately 30 seconds.
  Interventions: Other: Exercise; Other: Percussion massage therapy

INTERVENTIONS:
Other: Exercise — The exercise program will be performed at home twice daily for a period of four weeks. Participants will begin with 10 repetitions, and the number of repetitions will be individualized based on each person's clinical condition. They will be advised to discontinue any exercises that cause pain. An illustrated exercise brochure will be provided, and weekly follow-up will be conducted through phone calls to ensure adherence.
  At the start of the program, participants will be instructed to lie supine on a flat surface, bend their knees, and place approximately 30 cm of support (such as two pillows) under their lower legs to achieve a relaxation position, holding it for 30 seconds. The exercise program will include hip flexor and lumbar extensor stretching, hamstring stretching, bridge exercises, erector spinae strengthening in the prone "superman" position, quadruped alternating arm-leg lifts, and cat-camel exercises.
Other: IASTM — Instrument-assisted soft tissue mobilization will be administered twice a week for a total of eight sessions. The treatment will be performed using stainless steel tools of various sizes specifically designed for different anatomical regions. The intervention will target the iliocostalis lumborum, erector spinae, quadratus lumborum muscles, as well as both the superficial and deep fascia. Before beginning the procedure, a thin layer of petroleum jelly will be applied to the skin to ensure smooth gliding of the instrument.
  During the treatment, instrument-assisted mobilization will be applied over the muscle fibers using the sweep, fan, brush, and sweep techniques, with each technique performed for 8-10 repetitions. The total duration of the application will be six minutes.
  Arms: IASTM Group
Other: Percussion massage therapy — Vibration massage therapy will be administered twice per week for a total of eight sessions. After positioning the participant in the prone position, the treatment session will begin. The vibration massage will be delivered using the Theragun™ device equipped with the No. 2 standard ball attachment, operating at a frequency of 1750 percussions per minute. The device will be held perpendicular to the muscle throughout the application, and no additional pressure other than the weight of the device itself-will be applied. Continuous contact between the massage gun and the skin will be maintained to ensure consistent pressure. The intervention will target the erector spinae and lumbar paravertebral muscles. A total of 10 minutes of percussion massage will be applied to the lateral portions of the lower back, with 5 minutes administered to each side. During the treatment, the device will be guided in a straight path from the distal toward the proximal region within approximately 30 seconds.
  Arms: Percussion Massage Therapy Group

SUMMARY:
The aim of this study is to investigate the effects of Instrument-Assisted Soft Tissue Mobilization and vibration massage therapy on pain, functionality, and kinesiophobia in individuals with lumbar disc herniation.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of Instrument-Assisted Soft Tissue Mobilization and Percussion massage therapy on pain, functionality, and kinesiophobia in individuals with lumbar disc herniation. In addition, participants will be randomly assigned to three groups Conventional Therapy, Percussion Massage Therapy, and IASTM and the study will aim to examine and compare the pre- and post-treatment effects of these three interventions on pain, functionality, and kinesiophobia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 30 and 60 years of age
* Individuals diagnosed with lumbar disc herniation at the protrusion level
* Individuals with no cognitive, intellectual, or mental impairments and who are able to express themselves
* Individuals with a VAS score greater than 5
* Individuals experiencing pain for at least 3 months

Exclusion Criteria:

* Individuals with a history of lumbar surgery
* Individuals who are pregnant
* Individuals who have had a spinal tumor or any other malignancy within the past six months
* Individuals who have received physiotherapy for low back pain within the last six months
* Individuals with orthopedic conditions such as fractures
* Individuals diagnosed with neurological, rheumatological, or psychological disorders
* Individuals with diagnoses such as infection, spondylosis, spondylolysis, osteoporosis, or ankylosing spondylitis will be excluded from the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | From enrollment to the end of treatment at 4 weeks
  the Visual Analog Scale (VAS) will be used to assess pain intensity. VAS is a widely used tool in daily clinical practice for evaluating pain, and the average pain score ranges from 0 to 10. The VAS is typically defined as a 10-cm horizontal or vertical line that begins with "no pain" and ends with "unbearable pain." This line may be presented as a simple straight line or divided into equal segments. Participants will be asked to mark a point on the line that corresponds to the intensity of their pain. A score of "0" indicates no pain, scores of 1-4 represent mild pain, scores of 5-6 indicate moderate pain, and scores of 7-10 reflect severe pain.
Tampa Scale of Kinesiophobia | From enrollment to the end of treatment at 4 weeks
  The Tampa Scale of Kinesiophobia (TSK) will be used to assess kinesiophobia. This scale is commonly applied in individuals with acute and chronic low back pain, fibromyalgia, and musculoskeletal injuries. The TSK is a 17-item questionnaire developed to measure fear of movement and fear of reinjury, particularly in relation to work-related activities and fear-avoidance behaviors. It uses a 4-point Likert scoring system (1 = Strongly disagree, 4 = Strongly agree). The total score ranges from 17 to 68, with higher scores indicating greater levels of kinesiophobia.
The Oswestry Disability Index | From enrollment to the end of treatment at 4 weeks
  The Oswestry Disability Index (ODI) will be used to assess functional status. The ODI consists of 10 items scored on a scale from 0 to 5 and evaluates pain and limitations in various daily activities in individuals with low back pain. A score of 5 represents the highest level of disability for each item. The maximum possible score is 100%, indicating complete disability. The total score is interpreted across five categories: 0-20% reflects minimal disability, 21-40% indicates moderate disability, 41-60% represents severe disability, 61-80% corresponds to crippled patients, and 81-100% indicates individuals who are bedbound due to their condition.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Menek, Principal Investigator — Uludag University

IPD SHARING:
Plan to Share IPD: No